CLINICAL TRIAL: NCT06898515
Title: Fluid Management of Acute Decompensated Heart Failure Subjects Treated With Reprieve System (FASTR-II)
Brief Title: Fluid Management of Acute Decompensated Heart Failure Subjects Treated With Reprieve System (FASTR-II) (IDE-G210258)
Acronym: FASTR-II
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Reprieve Cardiovascular, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDE-G210258-CLN0002
Record Dates: First submitted 2025-03-10; First posted 2025-03-27 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Acute Decompensated Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Reprieve System (Experimental): Participants randomized to Reprieve System will receive personalized and optimized diuretic and saline infusion using the study device during the course of the treatment.
  Interventions: Device: Reprieve System
- Optimal Diuretic Therapy (ODT) (Active Comparator): Participants randomized to ODT will be treated with guided diuretic titration, as recommended in the ESC guidelines on diuretic therapy
  Interventions: Drug: furosemide infusion
- Registry (No Intervention): Participants will be treated per local site usual care.

INTERVENTIONS:
Device: Reprieve System — The Reprieve System is a hospital bedside fluid management console designed to provide personalized and automated infusion of the IV diuretic furosemide and physiological saline in response to the patient's real-time urine output to safely and rapidly decongest patients suffering from Acute Decompensated Heart Failure.
  Arms: Reprieve System
Drug: furosemide infusion — Participants randomized to ODT will be treated with guided diuretic titration, as recommended in the ESC guidelines on diuretic therapy
  Arms: Optimal Diuretic Therapy (ODT)

SUMMARY:
The objective of this study is to prospectively compare decongestive therapy administered by the Reprieve System to Optimal Diuretic Therapy (ODT) in the treatment of patients diagnosed with acute decompensated heart failure (ADHF). The main objective is to determine if the Reprieve System can more efficiently decongest ADHF patients in comparison to Control Therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HF with expected hospitalization >24 hours, with >1 new or worsening symptom and >2 physical examination, laboratory, or invasive findings of HF, and receiving or with plans to receive a HF-specific treatment
2. ≥10 lb. (4.5 kg) above dry weight as estimated by health care provider.
3. Current outpatient prescription for daily loop diuretic.
4. Participants ≥ 22 years of age able to provide informed consent and comply with study procedures.
5. Elevated risk of diuretic resistance, as indicated by at least one of the following: Baseline hypochloremia OR Urine output <1L in the 6 hours following IV loop diuretic >=40 mg furosemide equivalent OR Spot urine sodium <100 mmol/L 1-2 hours after IV loop diuretic >= 40 mg furosemide equivalent

Exclusion Criteria:

1. Urologic issues that would predispose the participant to a high rate of urogenital trauma or infection with catheter placement or known inability to place a Foley catheter.
2. Hemodynamic instability as defined by any of the following: sustained systolic blood pressure <90 mmHg for >15 minutes within the past 48 hours, use of IV vasopressors or inotropes within past 48 hours, and/or current or previous mechanical circulatory support within the last week.
3. Uncontrolled arrhythmias defined as sustained HR >130 beats/min for >10 minutes within the past 48 hours.
4. Severe lung disease with chronic home oxygen requirement >2L/min.
5. Acute infection with evidence of systemic involvement (e.g., clinically suspected infection with fever or elevated serum white blood cell count).
6. Estimated glomerular filtration rate (eGFR) <25 ml/min/1.73m2 (calculated with either MDRD or CKD-EPI) or current use of renal replacement therapy (RRT).
7. Significant left ventricular outflow obstruction, severe uncorrected complex congenital heart disease, known severe stenotic valvular disease, severe infiltrative or constrictive cardiomyopathy or other diagnosis that would make aggressive decongestion unsafe.
8. Current or recent (< 30 days) type I myocardial infarction (e.g., acute coronary syndrome such as NSTEMI or STEMI from plaque rupture), coronary artery bypass surgery, or stroke. An isolated troponin elevation (e.g., from volume overload or demand ischemia) is not a reason for exclusion.
9. Severe electrolyte abnormalities (e.g., serum potassium <3.0 mEq/L, magnesium <1.3 mEq/L or sodium <125 mEq/L). Note: These are based on baseline/screening labs. Participants whose electrolyte levels are repleted cannot be reassessed for inclusion in the trial.
10. Other concomitant disease or condition the investigator believes will make it difficult to follow instructions or comply with study procedures and/or follow-up visits, including expected prolonged hospitalization for reasons other than decongestive therapy
11. Currently enrolled in an interventional trial (observational studies are permitted).
12. Life expectancy less than 6 months.
13. Women who are pregnant or breastfeeding.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite/win-ratio | 1. up to 30 days from randomization, 2. up to 30 days from discharge, 3. up to 72 hours after randomization
  1. Freedom from 30-day CV mortality
  2. Freedom from HF Rehospitalization 30 days post-discharge
  3. Greater net sodium loss per 24 hours during treatment
Incidence of device/procedure-related adverse events (KDIGO stage 2 or greater AKI, CAUTI) | initiation of randomized therapy through 72 hours following completion of randomized therapy
  KDIGO stage 2 or greater AKI: ≥ doubling of serum creatinine or use of renal replacement therapy; CAUTI per CDC definition

SECONDARY OUTCOMES:
Net sodium loss | per 24 hours at end of randomized therapy
Time to discharge readiness | through hospital discharge, an average of 5 days
  Time from initiation of randomized therapy to when the participant becomes medically ready for discharge from a decompensated heart failure treatment standpoint
Time on IV diuretic therapy | randomization through hospital discharge, assessed up to 30 days
Net fluid loss | per 24 hours at end of randomized therapy
  Fluid input subtracted from total urine output
Weight loss | per 24 hours at end of randomized therapy
CV mortality and cumulative HF rehospitalizations | 90 days after hospital discharge
  Both types of events will be combined in a total "event rate" compared between groups
Length of stay | through hospital discharge, an average of 5 days
  Time from initiation of randomized therapy to hospital discharge
Hypotension defined as systolic blood pressure < 80 mmHg documented with two readings at least 30 minutes apart with symptoms (e.g., chest pain, dizziness) or <80 mmHg requiring an intervention including IV fluids or vasopressors. | initiation of randomized therapy up to 12 hours after stopping randomized therapy
Severe electrolyte abnormality | initiation of randomized therapy up to 72 hours after stopping randomized therapy
  serum potassium <3.0 mEq/L with ≥ 0.5 mEq/L decrease from initiation of randomized therapy, magnesium <1.3 mEq/L with ≥0.5 mEq/L decrease from initiation of randomized therapy, or sodium <125 mEq/L with ≥ 5.0 mEq/L decrease from initiation of randomized therapy
Worsening heart failure requiring a higher level of HF therapy | initiation of randomized therapy up to 72 hours after stopping randomized therapy
Tinnitus or hearing loss lasting more than 30 minutes | initiation of randomized therapy up to 12 hours after stopping randomized therapy

CONTACTS AND LOCATIONS:
Overall Officials: Javed Butler, MD, MPH, MBA, Principal Investigator — Baylor Scott and White Health
Locations (53):
- United States (37):
  - University of California Irvine, Irvine, California
  - Scripps Memorial Hospital, La Jolla, California
  - UC Davis Medical Center, Sacramento, California
  - University of Florida, Gainesville, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Piedmont Augusta Hospital, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville Hospital, Louisville, Kentucky
  - Trinity Health Ann Arbor Hospital, Ann Arbor, Michigan
  - Corewell Health Butterworth Hospital, Grand Rapids, Michigan
  - Corewell William Beaumont University Hospital, Royal Oak, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Mississippi, Jackson, Mississippi
  - Harry S. Truman Veteran's Memorial Hospital, Columbia, Missouri
  - St. Louis VA, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Stony Brook University Hospital, Stony Brook, New York
  - Duke University, Durham, North Carolina
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Lindner Center at Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - UH Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Baylor Scott and White, Dallas, Texas
  - Baylor College of Medicine Ben Taub Hospital, Houston, Texas
  - Memorial Hermann-Texas Medical Center, Houston, Texas
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - VCU Medical Center, Richmond, Virginia
  - UW Harborview, Seattle, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Germany (4):
  - Universitätsklinikum Gießen (UKGM), Giessen
  - Hannover University Hospital, Hanover
  - University Hospital Heidelberg, Heidelberg
  - Jena University Hospital, Jena
- Italy (3):
  - Universitaria delle Marche, Ancona
  - ASST Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - ASST Niguarda Great Metropolitan Hospital, Milan
- Poland (3):
  - Medical University of Białystok, Bialystok
  - Medical University of Lodz, Lodz
  - University Hospital Wroclaw, Wroclaw
- Spain (6):
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital de Bellvitge, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Puerta de Hierro Majadahonda University Hospital, Madrid
  - Clínico Universitario de Valencia, Valencia
  - Hospital General Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No